CLINICAL TRIAL: NCT06978036
Title: Single-blinded Randomized Non-inferiority Controlled Clinical Trial Comparing Endoscope-assisted Flapless Approach Versus Papillary Preservation Technique in Periodontal Regeneration of Intra-bony Periodontal Defects
Brief Title: Endoscope-assisted Flapless Approach Versus Papillary Preservation Technique in Periodontal Regeneration.
Acronym: EAFAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Melissa Fok, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P&ID2025_02
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis; Periodontal Regeneration, Clinical and Radiographic Results, Modified Minimal Invasive Surgery; Periodontal Regeneration
Keywords: Periodontitis; Intrabondy defects; Perioscope; Perioscopy; endoscope-assisted; regeneration; papilla preservation; enamel matrix derivative
MeSH Terms: conditions — Periodontitis | interventions — emerin

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized non-inferiority controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flapless EASD + EMD (Experimental): Periodontal regneration with EMD in conjuction with Endoscope-assisted subgingival debridement
  Interventions: Procedure: Flapless periodontal regeneration with EMD + EASD
- PPT + EMD (Active Comparator): Periodontal regneration with periodontal surgery using Papilla Presevation Technique
  Interventions: Procedure: Periodontal regeneration with EMD + PPT

INTERVENTIONS:
Procedure: Flapless periodontal regeneration with EMD + EASD — Periodontal regneration with EMD in conjuction with Endoscope-assisted subgingival debridement
  Arms: Flapless EASD + EMD
Procedure: Periodontal regeneration with EMD + PPT — Periodontal regneration with EMD in conjunction with periodontal surgery using Papilla Presevation Technique
  Arms: PPT + EMD

SUMMARY:
The standard of care for regeneration of lost periodontal tissue from disease at contained defect sites non-responding to non-surgical periodontal therapy is periodontal regenerative surgery. The classical practice of periodontal regeneration involves an open flap surgical approach with the the application of biologics (Enamel matrix derivatives EMD) and biomaterials after root surface debridement. EMD, derived from porcine, has been well documented for its safety and efficacy and widely used in periodontal regeneration. There is some evidence demonstrating promising treatment outcome of the flapless application of periodontal regenerative biologics after nonsurgical subgingival debridement. Endoscopic-Assisted Subgingival Debridement EASD with a high magnification up to 40X has been shown to be a non-inferior nonsurgical treatment alternative to open flap debridement with shorter operation times and better early wound healing. We hypothesize that EASD could be integrated into flapless periodontal regeneration to improve clinical performance, patient comfort and acceptance to regenerative procedures. Hence, the focus of this study is to investigate whether flapless application of EMD as an adjunct to EASD can achieve non-inferior clinical results compared to classical open-flap periodontal regeneration using Papilla Preservation Surgical Technique PPT in managing residual periodontal intrabony defects 1 year after intervention. Half of the patients will be randomized to recieve EASD and flapless regneration with EMD, while the other half of the patient will receive classical regeneration with PPT and EMD.

ELIGIBILITY:
Inclusion Criteria:

* Stage III - Stage IV Periodontitis patients, 3-4 months after completing steps I & II periodontal therapy.
* At least 1 tooth presented with 1 site with >5mm residual PPD and ≥6mm CAL, with ≥3mm intra-osseous defect presented involving predominantly the interdental space of the tooth and presented on paralleling periapical radiographs and/or CBCT.
* Presence of a periodontally stable tooth with PPD≤3mm immediate adjacent to the intra-bony defect of the investigated tooth
* Good Oral Hygiene, with Full Mouth Plaque Score ≤25% at baseline and with good plaque control at proposed surgical field.

Exclusion Criteria:

* Pre-study period

  * Any systemic condition which prevents following the study protocol;
  * Any systemic condition which may affect healing outcomes of patients, e.g. uncontrolled or poorly controlled diabetes, unstable or life-threatening conditions or those requiring antibiotic prophylaxis;
  * Patients under long-term analgesic medication;
  * Current smokers;
  * Self-reported pregnancy;
  * Systemic antimicrobial therapy within 3 months;
  * Teeth that concurrently present with a buccal and a lingual intrabony defect component;
  * Tooth with hopeless prognosis or questionable prognosis associated with endodontic lesions, or subgingival restorations that preclude clinical measurements, or excessive uncontrolled mobility;
  * Any factors which prohibit regular performance of plaque control around surgical sites;
  * Inadeduate oral hygiene with full mouth plaque score >25%
  * Furcation involved surfaces
* During study period -Non-compliance with study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
ΔCAL - 12 months | 12 months
  Change of Clinical Attachment Level measured in millimetres

SECONDARY OUTCOMES:
ΔCAL - 6 months | 6 months
  Change of Clinical Attachment Level, measured in milimetres
ΔCAL - 9 months | 9 months
  Change of Clinical Attachment Level, measured in milimetres
FMPS | 3, 6, 9, 12 months
  Modified O'Leary Full Mouth Plaque Score, measured in percentage
FMBOP | 3, 6, 9, 12 months
  Full Mouth Bleeding On Probing (excluding teeth under investigation), measured in percentage
ΔREC | 3, 6, 9, 12 months
  Change in Recession , measured in milimetres
ΔPPD | 6, 9, 12 months
  Change in Periodontal Pocket Depth, measrued in millimetres
Mob | 3, 6, 9, 12 months
  Tooth Mobility Index (Miller 1938), the higher the number the greater the mobility
EWHI | 3, 6, 9, 12 months
  Early Wound Healing Index (Wachtel et al., 2003), a lower score signifies a better healing
ΔINFRA | 3, 6, 9, 12 months
  Change of depth of the intrabony defect , measured on radiographs in millimetres.
TIME | Measured throughout procedure
  Time for the surgery , measured in minutes
% of sites achieving therapeutic endpoints | 6, 9, 12 months
  % of sites achieving therapeutic endpoints (i.e. no PPD > 4mm with bleeding and no deep residual pocket PPD >5mm)
Patient-reported outcome measurements | Baseline, 3, 6, 9, 12 months
  Subjects will be assessed with a questionnaire on condition-specific Health-related quality-of-life instrument and perceptions of oral health-related quality of life will be assessed using validated translations of the OHIP-14 questionnaire into the native language of all participants. A lower value indicates a more favourable patient-reported outcome.
Intra-operative Discomfort | 14 days
  100mm Visual Analog Scale is used to measure the intra-operative pain and discomfort during the test/control therapy.
Daily intake of analgesia | 14 days
  Daily intake of analgesia will be recorded on the first 14 days after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is concern that individual participant data sharing may violate data ownership policy of the institute. Information sheet and consent form approved by local IRB did not explicitly permit data sharing beyond the scope of the current study. As such, sharing IPD could potentially infringe upon the rights and expectations of our participants, which we are committed to safeguarding.